CLINICAL TRIAL: NCT00959894
Title: Antiretroviral Activity and Tolerability of Once Daily Etravirine in Treatment-Naïve Adults With HIV-1 Infection
Brief Title: Evaluating Once Daily Etravirine in Treatment-Naive Adults With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Michelle Floris-Moore, MD, Clinical Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-2070
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: HIV Infections
Keywords: HIV; Infection; Treatment Naive; Adults; Once; Daily; Etravirine; HIV-1 Infection
MeSH Terms: conditions — HIV Infections; Infections | interventions — etravirine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etravirine 400 mg once daily (Experimental): Etravirine 400 mg once daily with fixed dose tenofovir/emtricitabine (Truvada) one tablet once daily
  Interventions: Drug: Etravirine (Intelence); Drug: Truvada

INTERVENTIONS:
Drug: Etravirine (Intelence) — Etravirine 400 mg (four 100 mg or two 200 mg tablets) taken orally once a day with one pill of Truvada (200 mg of emtricitabine and 300 mg of tenofovir) taken orally once a day
  Other Names: TMC-125; Intelence
Drug: Truvada — Etravirine 400 mg (four 100 mg or two 200 mg tablets) taken orally once a day with one pill of Truvada (200 mg of emtricitabine and 300 mg of tenofovir) taken orally once a day
  Other Names: Tenofovir/emtricitabine

SUMMARY:
The main study is a single arm, open-label, prospective study to assess antiretroviral activity and tolerability of etravirine (TMC-125) 400 mg once daily, given with fixed-dose tenofovir/emtricitabine, in treatment-naïve HIV-1-infected men and women. There are also a genital secretions pharmacokinetic (PK) sub-study and a metabolic sub-study. The purpose of the genital secretions PK sub-study is to gain information about drug levels and HIV-1 RNA in genital secretions when subjects are taking etravirine. The purpose of the metabolic sub-study is to learn about the effects of etravirine on body composition, as well as lipid and glucose levels.

DETAILED DESCRIPTION:
Participants: There will be approximately 80 HIV-1-infected men and women aged 18 years or older who have taken less than or equal to 10 days of prior antiretroviral therapy and have never taken etravirine, dapivirine (TMC120), or rilpivirine (TMC 278) in the main study. There will be approximately 40 subjects who enroll in the main study that will be in the metabolic sub-study and approximately 20 subjects (10 pre-menopausal women and 10 men) who enroll in the main study that will be in the genital secretions PK sub-study.

Procedures (methods): For the main study subjects will take etravirine 400 mg once daily orally with fixed-dose tenofovir/emtricitabine (Truvada) one tablet once daily. For the genital secretions PK sub-study, genital secretion samples will be self-collected throughout the study except for the week 4 study visit where women will have the cervicovaginal sample at time 0 and at 24 hours collected by study staff. For the metabolic sub-study, waist measurements and dual energy x-ray absorptiometry (DEXA) scans will be performed at entry, week 24, and week 96, and 2-3 teaspoons of blood to check lipids, insulin, and glucose will be taken at entry and weeks 12, 24, 48, and 96.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by any licensed ELISA test and confirmed by Western Blot or other confirmatory test at any time prior to study entry. Acceptable alternative confirmatory tests are plasma HIV-1 RNA, HIV-1 culture, HIV-1 antigen, or a second antibody test by a method other than ELISA. Alternatively, if an HIV-antibody test result is not available, two HIV-1 RNA values >2000 copies/mL, drawn at least 24 hours apart, performed by any laboratory that has clinical laboratory improvement amendments (CLIA) certification, or its equivalent, may be used to document infection.
* Age 18 years or older.
* Able to provide informed consent.
* In the opinion of the investigator, able to comply with study medication and procedures.
* Plasma HIV-1 RNA ≥ 1000 copies/mL as measured by any FDA-approved test for quantifying HIV-1 RNA within 90 days prior to study entry.
* Less than or equal to 10 days of cumulative exposure to antiretroviral therapy.
* For all women of reproductive potential, a negative urine or serum β-human chorionic gonadotropin (β-HCG) pregnancy test performed within 48 hours prior to study entry.

  * All study volunteers, both male and female, must agree not to participate in a conception process (i.e., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) while receiving study medications and for 6 weeks after stopping study medications.
  * If participating in sexual activity that could lead to conception, study volunteers must agree to use at least one method of reliable contraception which must be a barrier method (i.e., a condom without spermicide, a diaphragm, or cervical cap) throughout the study and for 6 weeks thereafter.

NOTE: Acceptable documentation of lack of reproductive potential for a woman is self-reported history of being postmenopausal for at least 24 months, or having had surgical sterilization (hysterectomy, or bilateral oophorectomy, or bilateral tubal ligation) or of male partner's azoospermia. Acceptable documentation for a man is self-reported history of azoospermia.

* Hemoglobin ≥ 7.5 g/dL within 45 days prior to study entry.
* Absolute neutrophil count ≥ 500/mm³ within 45 days prior to study entry.
* Platelets ≥ 50,000/mm³ within 45 days prior to study entry.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3X upper limit of normal (ULN) or bilirubin ≤ 2.5 ULN within 45 days prior to study entry.
* Glomerular filtration rate (GFR) > 59 as calculated by Modification of Diet in Renal Disease (MDRD) equation within 45 days prior to study entry.

Exclusion Criteria:

* Prior receipt of etravirine, dapivirine, or rilpivirine (Edurant), or Complera.
* Evidence of any of the resistance-associated mutations listed below on genotype testing performed within 90 days of study entry. Any pending resistance testing ordered prior to study entry must be available for review by the investigator prior to enrollment. Major resistance mutations include:

  1. Any of the following nonnucleoside reverse transcriptase inhibitor (NNRTI) mutations: V90I, A98G, L100I, K101E/H/P/Q, K103H/S/T, V106A/I/M, V108I, E138A/G/K/Q, V179D/E/F/G/I/T, Y181C/I/V, Y188C/H/L, V189I, G190A/C/E/Q/S, H221Y, P225H, F227C/L, M230I/L, P236L, K238N/T, K103N.
  2. Any of the following NRTI mutations: M184V/I, K70E/R, K65R, M41L, 69 insert, L210W, T215Y/F, K219Q/E, L74V.
* Pregnancy
* Breastfeeding
* Any condition which, in the opinion of the investigator, would be likely to interfere with ability to take the study medications appropriately and comply with the study protocol.
* Use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 30 days prior to study entry.

NOTE: Routine standard of care, including hepatitis B, influenza, pneumococcus, and tetanus vaccines are permitted.

* Current active illness requiring systemic treatment and/or hospitalization until the individual completes therapy or, in the opinion of the investigator, is clinically stable on therapy for at least 7 days prior to study entry.
* Life expectancy of less than 6 months.
* Acute viral hepatitis.
* Known allergy/hypersensitivity to components of the study drugs or their formulations.
* Use of any medications that are prohibited during the study period (see Section 8.1 of the protocol - Prohibited Medications).
* Refusal by an individual who is taking anti-depressant medications to allow the investigator or Primary HIV Care provider to communicate with his/her psychiatrist/Mental Health clinician regarding the initiation of study medications in those cases where co-administration of study drugs may alter anti-depressant drug levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Floris-Moore, MD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

REFERENCES:
- [Background] Gruzdev B, Rakhmanova A, Doubovskaya E, Yakovlev A, Peeters M, Rinehart A, de Dier K, Baede-Van Dijk P, Parys W, van 't Klooster G. A randomized, double-blind, placebo-controlled trial of TMC125 as 7-day monotherapy in antiretroviral naive, HIV-1 infected subjects. AIDS. 2003 Nov 21;17(17):2487-94. doi: 10.1097/00002030-200311210-00011. PMID 14600520
- [Background] TMC125-C223 Writing Group; Nadler JP, Berger DS, Blick G, Cimoch PJ, Cohen CJ, Greenberg RN, Hicks CB, Hoetelmans RM, Iveson KJ, Jayaweera DS, Mills AM, Peeters MP, Ruane PJ, Shalit P, Schrader SR, Smith SM, Steinhart CR, Thompson M, Vingerhoets JH, Voorspoels E, Ward D, Woodfall B. Efficacy and safety of etravirine (TMC125) in patients with highly resistant HIV-1: primary 24-week analysis. AIDS. 2007 Mar 30;21(6):F1-10. doi: 10.1097/QAD.0b013e32805e8776. PMID 17413684
- [Background] Shikuma CM, Yang Y, Glesby MJ, Meyer WA 3rd, Tashima KT, Ribaudo HJ, Webb N, Bastow B, Kuritzkes DR, Gulick RM. Metabolic effects of protease inhibitor-sparing antiretroviral regimens given as initial treatment of HIV-1 Infection (AIDS Clinical Trials Group Study A5095). J Acquir Immune Defic Syndr. 2007 Apr 15;44(5):540-50. doi: 10.1097/QAI.0b013e318031d5a0. PMID 17245230
- [Background] Madruga JV, Cahn P, Grinsztejn B, Haubrich R, Lalezari J, Mills A, Pialoux G, Wilkin T, Peeters M, Vingerhoets J, de Smedt G, Leopold L, Trefiglio R, Woodfall B; DUET-1 study group. Efficacy and safety of TMC125 (etravirine) in treatment-experienced HIV-1-infected patients in DUET-1: 24-week results from a randomised, double-blind, placebo-controlled trial. Lancet. 2007 Jul 7;370(9581):29-38. doi: 10.1016/S0140-6736(07)61047-2. PMID 17617270
- [Background] Lazzarin A, Campbell T, Clotet B, Johnson M, Katlama C, Moll A, Towner W, Trottier B, Peeters M, Vingerhoets J, de Smedt G, Baeten B, Beets G, Sinha R, Woodfall B; DUET-2 study group. Efficacy and safety of TMC125 (etravirine) in treatment-experienced HIV-1-infected patients in DUET-2: 24-week results from a randomised, double-blind, placebo-controlled trial. Lancet. 2007 Jul 7;370(9581):39-48. doi: 10.1016/S0140-6736(07)61048-4. PMID 17617271
- [Background] Ghosn J, Chaix ML, Peytavin G, Rey E, Bresson JL, Goujard C, Katlama C, Viard JP, Treluyer JM, Rouzioux C. Penetration of enfuvirtide, tenofovir, efavirenz, and protease inhibitors in the genital tract of HIV-1-infected men. AIDS. 2004 Sep 24;18(14):1958-61. doi: 10.1097/00002030-200409240-00014. PMID 15353984
- [Background] Reddy YS, Gotzkowsky SK, Eron JJ, Kim JY, Fiske WD, Fiscus SA, Petch L, Cohen MS, Kashuba AD. Pharmacokinetic and pharmacodynamic investigation of efavirenz in the semen and blood of human immunodeficiency virus type 1-infected men. J Infect Dis. 2002 Nov 1;186(9):1339-43. doi: 10.1086/344311. Epub 2002 Oct 7. PMID 12402205
- [Background] Taylor S, Reynolds H, Sabin CA, Drake SM, White DJ, Back DJ, Pillay D. Penetration of efavirenz into the male genital tract: drug concentrations and antiviral activity in semen and blood of HIV-1-infected men. AIDS. 2001 Oct 19;15(15):2051-3. doi: 10.1097/00002030-200110190-00022. PMID 11600838
- [Background] van Praag RM, Repping S, de Vries JW, Lange JM, Hoetelmans RM, Prins JM. Pharmacokinetic profiles of nevirapine and indinavir in various fractions of seminal plasma. Antimicrob Agents Chemother. 2001 Oct;45(10):2902-7. doi: 10.1128/AAC.45.10.2902-2907.2001. PMID 11557488
- [Background] Scholler-Gyure M, Kakuda TN, De Smedt G, Woodfall B, Lachaert R, Beets G, Peeters M, Hoetelmans RM. Pharmacokinetics of TMC125 in once- and twice- daily regimens in HIV-1-negative volunteers. Program and Abstracts of the 47th Interscience Conference on Antimicrobial Agents and Chemotherapy, 2007 [Abstract A-1427], Chicago IL.
- [Background] Lalezari J, et al. Pharmacokinetics of once-daily etravirine (ETR) without and with once-daily darunavir/ritonavir (DRV/r) in antiretroviral-naïve HIV-1 infected adults. 9th International Congress on Drug Therapy in HIV Infection 2008; abstract O413.
- [Background] 144-week data released on Gilead's study 934. AIDS Patient Care STDS. 2007 Aug;21(8):603-4. No abstract available. PMID 17902243
- [Derived] Floris-Moore MA, Mollan K, Wilkin AM, Johnson MA, Kashuba AD, Wohl DA, Patterson KB, Francis O, Kronk C, Eron JJ. Antiretroviral activity and safety of once-daily etravirine in treatment-naive HIV-infected adults: 48-week results. Antivir Ther. 2016;21(1):55-64. doi: 10.3851/IMP2982. Epub 2015 Aug 11. PMID 26263403

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 80 participants were enrolled, however 1 participant was found to be ineligible on the day of entry and never started study medication (had developed acute renal failure and therefore no longer met eligibility requirements).
Period: Overall Study
Arm/Group | Etravirine 400 mg Once Daily
Started | 79 (One (1) additional subject became ineligible on the day of entry and never started study medication.)
Completed | 63
Not Completed | 16
Not completed — Lost to Follow-up | 10
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Need for contraindicated medication | 1
Not completed — Subject moved out of town | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study medication (etravirine 400 mg given once daily with with one tablet of fixed dose tenofovir/emtricitabine).
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [23 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 71
Region of Enrollment [Number; unit: participants]
  United States | 79

OUTCOME MEASURES:

1. Primary Outcome: The Antiretroviral Activity of Etravirine 400 mg Given Once Daily, With Fixed-dose Truvada Once Daily, Among Treatment-naïve HIV-1 Infected Adults as Measured by the Percentage of Participants With HIV RNA < 50 Copies/mL at Week 24
Description: The primary study endpoint was the proportion of participants who achieved HIV-1 RNA <50 copies/ml at Week 24 of study participation. The per-protocol primary analysis was conducted intention-to-treat, with missing evaluations counted as failures. Achievement of HIV-1 viral load below 50 copies/ml was defined as having HIV-1 RNA <50 copies/ml during the Week 24 analysis window (>18 and <30 weeks post-entry).
Time Frame: 24 weeks
Population: Of 79 participants who initiated study medications, 74 had a Week 24 HIV-1 RNA measurement. The primary analysis was conducted intention-to-treat, with missing evaluations counted as failure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.87 [0.78 to 0.94]

2. Secondary Outcome: The Proportion of Participants With HIV RNA <50 Copies/mL at Week 48 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: This secondary outcome assessed the proportion of participants who achieved HIV-1 RNA <50 copies/ml at Week 48 of study treatment. The per-protocol analysis was conducted intention-to-treat, with missing evaluations counted as failures.
Time Frame: 48 weeks
Population: Of 79 participants who initiated study medications, 69 had a Week 48 HIV-1 RNA measurement (4 participants had discontinued the study, 3 were lost to follow-up, and 3 missed the Week 48 visit). The analysis was conducted intention-to-treat, with missing evaluations counted as failure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.77 [0.66 to 0.86]

3. Secondary Outcome: The Proportion of Participants With HIV RNA <50 Copies/mL at Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: This secondary outcome assessed the proportion of participants who achieved HIV-1 RNA <50 copies/ml at Week 96 of study treatment. The per-protocol analysis was conducted intention-to-treat, with missing evaluations counted as failures.
Time Frame: 96 weeks
Population: Of 79 participants who initiated study medications, 63 had a Week 96 HIV-1 RNA measurement (6 participants had discontinued the study and 10 were lost to follow-up). The analysis was conducted intention-to-treat, with missing evaluations counted as failure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.71 [0.60 to 0.81]

4. Secondary Outcome: The Proportion of Participants With HIV RNA <200 Copies/mL at Week 24 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: This secondary outcome assessed the proportion of participants who achieved HIV-1 RNA <200 copies/ml at Week 24 of study treatment. The per-protocol analysis was conducted intention-to-treat, with missing evaluations counted as failures.
Time Frame: 24 weeks
Population: Of 79 participants who initiated study medications, 74 had a Week 24 HIV-1 RNA measurement (3 participants had discontinued the study, 1 was lost to follow-up, and 1 missed the Week 24 visit). The analysis was conducted intention-to-treat, with missing evaluations counted as failure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.89 [0.79 to 0.95]

5. Secondary Outcome: The Proportion of Participants With HIV RNA <200 Copies/mL at Week 48 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: This secondary outcome assessed the proportion of participants who achieved HIV-1 RNA <200 copies/ml at Week 48 of study treatment. The per-protocol analysis was conducted intention-to-treat, with missing evaluations counted as failures.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.82 [0.72 to 0.90]

6. Secondary Outcome: The Proportion of Participants With HIV RNA <200 Copies/mL at Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: This secondary outcome assessed the proportion of participants who achieved HIV-1 RNA 200 copies/ml at Week 96 of study treatment. The per-protocol analysis was conducted intention-to-treat, with missing evaluations counted as failures.
Time Frame: 96 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.77 [0.66 to 0.86]

7. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 24 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: The per-protocol analysis of change in CD4+ cell count from baseline to Week 24 was calculated using the measurement closest to schedule and within the analysis window, and quantified with an estimated median and distribution-free 95% confidence interval (CI).
Time Frame: Baseline to 24 weeks
Population: Of 79 participants who initiated study medications, 73 had a Week 24 CD4+ cell count measurement (4 discontinued study participation prior to Week 24,1 missed the Week 24 visit, and 1 did not have a Week 24 CD4+ cell count measurement).
Measure: Median (95% Confidence Interval); unit: cells/uL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 73
cells/uL | 156 [113 to 200]

8. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 48 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: The per-protocol intention-to-treat analysis of change in CD4+ cell count from baseline to Week 48 was calculated using the measurement closest to schedule and within the analysis window, and quantified with an estimated median and distribution-free 95% CI.
Time Frame: Baseline to 48 weeks
Population: Of 79 participants who initiated study medications, 69 had a Week 48 CD4+ cell count measurement (4 discontinued study participation prior to Week 48 visit, 3 were lost to follow-up, and 3 missed the Week 48 visit).
Measure: Median (95% Confidence Interval); unit: cells/uL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 69
cells/uL | 163 [136 to 203]

9. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: The per-protocol intention-to-treat analysis of change in CD4+ cell count from baseline to Week 96 was calculated using the measurement closest to schedule and within the analysis window, and quantified with an estimated median and distribution-free 95% CI.
Time Frame: Baseline to 96 weeks
Population: Of 79 participants who initiated study medications, 63 had a Week 48 CD4+ cell count measurement (6 discontinued study participation prior to Week 96 and 10 were lost to follow-up).
Measure: Median (95% Confidence Interval); unit: cells/uL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 63
cells/uL | 224 [188 to 266]

10. Secondary Outcome: Resistance Mutations in the Subset of Patients With Confirmed Virologic Failure Who Have HIV RNA >500 Copies/mL and Genotype Resistance Results
Description: Per-protocol, genotype testing was conducted at confirmation of virologic failure if the confirmatory HIV-1 RNA was above the laboratory-specified threshold of 500 copies/mL. HIV-1 genotype was determined using the TRUGENE® HIV-1 assay (Siemens Healthcare Diagnostics, Tarrytown, NY)
Time Frame: 96 weeks
Population: Of participants with confirmed virologic failure, 8 had HIV-1 RNA levels ≥ 500 copies/mL and 6 of these had viral genotype results available (1 had previously discontinued study medication at Week 2, and 1 was missing).
Measure: Number; unit: participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 6
participants
  Y181C | 1
  E138K | 1
  E138K, Y181C, M230L, M184I, K219E, V75I | 1
  No resistance-associated mutations detected | 3

11. Secondary Outcome: Tolerability of Etravirine in HIV-1 Infected Adults Initiating Antiretroviral Therapy
Description: The safety/tolerability endpoint was defined as the first grade 3 or higher sign, symptom or laboratory abnormality that was at least one grade higher than baseline among participants ever exposed to etravirine (regardless of treatment status), or permanent discontinuation of etravirine due to any toxicity (regardless of grade). Modification of tenofovir/emtricitabine was not a safety/tolerability event.
  The Kaplan-Meier method was used to estimate the proportion of participants ever exposed to etravirine who remained event-free through Week 96, with a 95% CI using Greenwood's variance estimate and a log-log transformation. Time was handled as continuous (weeks from treatment start to event or censoring).
Time Frame: 96 weeks
Population: The analysis population for this outcome is all participants who received at least one dose of etravirine, regardless of whether or not they were still receiving etravirine at the time of the safety/tolerability event.
Measure: Number; unit: participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
participants
  At least one safety/tolerability event | 23
  Signs or Symptoms | 13
  Laboratory Abnormalities | 10

12. Secondary Outcome: Probability of Remaining Free of a Safety/Tolerability Event at 96 Weeks
Description: The Kaplan-Meier method was used to estimate the proportion of participants ever exposed to etravirine who remained event-free through Week 96, with a 95% CI using Greenwood's variance estimate and a log-log transformation. Time was handled as continuous (weeks from treatment start to event or censoring).
Time Frame: 96 weeks
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 79
proportion of participants | 0.69 [0.57 to 0.78]

13. Secondary Outcome: Change in the Lipid Profile and Glucose Metabolism, in a Subgroup of up to 40 Participants, From Baseline to Week 24 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: Metabolic data analyses were conducted as-treated. Changes in total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, triglycerides, and fasting blood glucose from baseline to follow-up were calculated using the value closest to schedule and within the analysis window, and were quantified with the median and inter-quartile range.
Time Frame: Baseline to 24 weeks
Population: This per-protocol sub-study analysis of metabolic outcomes was conducted in the as-treated population in the metabolic sub-study.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 36
mg/dL
  Total cholesterol | -7 [-17 to 4]
  HDL-cholesterol | 1 [-4 to 9]
  LDL-cholesterol | -9 [-14 to -1]
  Triglycerides | -16 [-33 to 18]
  Fasting glucose | 1 [-6 to 9]

14. Secondary Outcome: Change in Glucose Metabolism (Insulin Resistance), in a Subgroup of up to 40 Participants, From Baseline to Week 24 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: Metabolic data analyses were conducted as-treated. Insulin resistance was estimated by the homeostasis model assessment of insulin resistance (HOMA-IR), and was calculated as [fasting insulin (µU/mL) × fasting glucose (mmol/L)]/22.5. Changes from baseline to follow-up were calculated using the value closest to schedule and within the analysis window, and were quantified with the median and inter-quartile range.
Time Frame: Baseline to 24 weeks
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: µU/ml*mmol/L
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 27
µU/ml*mmol/L | -0.08 [-0.72 to 0.27]

15. Secondary Outcome: Change in the Lipid Profile and Glucose Metabolism, in a Subgroup of up to 40 Participants, From Baseline to Week 48 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: as for outcome 13
Time Frame: Baseline to 48 weeks
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 32
mg/dL
  Total cholesterol | 6 [-14 to 21]
  HDL-cholesterol | 5 [-2 to 12]
  LDL-cholesterol | -1 [-10 to 14]
  Triglycerides | -10 [-26 to 21]
  Fasting glucose | 2 [-5 to 6]

16. Secondary Outcome: Change in Glucose Metabolism (Insulin Resistance), in a Subgroup of up to 40 Participants, From Baseline to Week 48 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: as for outcome 14
Time Frame: Baseline to 48 weeks
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: µU/ml*mmol/L
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 23
µU/ml*mmol/L | 0.71 [-0.01 to 2.21]

17. Secondary Outcome: Change in the Lipid Profile and Glucose Metabolism, in a Subgroup of up to 40 Participants, From Baseline to Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: Metabolic data analyses were conducted as-treated. Changes in total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, triglycerides, and fasting blood glucose from baseline to follow-up were calculated using the value closest to schedule and within the analysis window, and were quantified with the median and inter-quartile range. Insulin resistance was estimated by the homeostasis model assessment of insulin resistance (HOMA-IR), and was calculated as [fasting insulin (µU/mL) × fasting glucose (mmol/L)]/22.5.
Time Frame: Baseline to 96 weeks
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 22
mg/dL
  Total cholesterol | 6 [-14 to 21]
  HDL-cholesterol | 4 [-3 to 15]
  LDL-cholesterol | -5 [-26 to 7]
  Triglycerides | 3 [-18 to 16]
  Fasting glucose | 2 [-6 to 6]

18. Secondary Outcome: Change in Glucose Metabolism (Insulin Resistance), in a Subgroup of up to 40 Participants, From Baseline to Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: as for outcome 14
Time Frame: Baseline to 96 weeks
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: µU/ml*mmol/L
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 18
µU/ml*mmol/L | 0.23 [-0.67 to 1.15]

19. Secondary Outcome: Change in Limb and Trunk Fat Distribution as Measured by DEXA Scan, in the Same Subgroup of up to 40 Participants (as in Aim 8), From Baseline to Week 24 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: Changes from baseline to follow-up in limb fat, trunk fat, total body fat, and lean mass were calculated. Whole body Dual X-ray Absorptiometry (DEXA) scans (Hologic Discovery W, Hologic Inc., Bedford, MA) were conducted at baseline, Week 24, and Week 96 to assess body fat distribution. Calculations of change from baseline to follow-up used the value closest to schedule and within the analysis window, and were quantified with the estimated median and distribution-free 95% CI.
Time Frame: Baseline to 24 weeks
Population: This per-protocol sub-study analysis was conducted in the as-treated population of participants in the metabolic sub-study.
Measure: Median (95% Confidence Interval); unit: percentage of body fat
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 37
percentage of body fat
  Total body fat | 0.43 [-0.63 to 1.10]
  Limb fat | 0.48 [-0.64 to 0.99]
  Trunk fat | 0.32 [-0.41 to 1.66]

20. Secondary Outcome: Change in Limb and Trunk Fat Distribution as Measured by DEXA Scan, in the Same Subgroup of up to 40 Participants (as in Aim 8), From Baseline to Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: as for outcome 19
Time Frame: Baseline to 96 weeks
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: percentage of body fat
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 25
percentage of body fat
  Total body fat | 1.44 [-0.40 to 3.86]
  Limb fat | 0.82 [-1.55 to 4.12]
  Trunk fat | 1.93 [0.31 to 4.67]

21. Secondary Outcome: Change in Fat Mass Ratio as Measured by DEXA Scan, in the Same Subgroup of up to 40 Participants (as in Aim 8), From Baseline to Week 24 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: Change from baseline to follow-up in fat mass ratio was calculated. Whole body Dual X-ray Absorptiometry (DEXA) scans (Hologic Discovery W, Hologic Inc., Bedford, MA) were conducted at baseline, Week 24, and Week 96 to assess body fat distribution. Fat mass ratio was calculated as the ratio of trunk fat percentage and lower limb fat percentage (% trunk fat mass / % lower limb fat mass). Calculations of change from baseline to follow-up used the value closest to schedule and within the analysis window, and were quantified with the estimated median and distribution-free 95% CI.
Time Frame: Baseline to 24 weeks
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: ratio of trunk fat % : lower limb fat %
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 37
ratio of trunk fat % : lower limb fat % | 0.02 [-0.01 to 0.09]

22. Secondary Outcome: Pharmacokinetics of Etravirine in Genital Secretions of up to 10 Men and up to 10 Women at Week 4 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: This secondary outcome measure assessed the ratio of semen:plasma concentration of etravirine in paired semen and plasma samples collected from 14 male participants at Week 4 of treatment with etravirine and fixed dose tenofovir/emtricitabine.
Time Frame: 4 weeks
Population: Of 79 participants who initiated study medications, 14 provided paired plasma and genital secretion samples. The goal was to enroll a total of 20 participants (10 men and 10 women) into the genital secretion sub-group, however no women enrolled into this subgroup. Data are presented for semen and plasma etravirine concentrations for 14 men.
Measure: Median (Inter-Quartile Range); unit: ratio of semen:plasma drug concentration
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 14
ratio of semen:plasma drug concentration | 0.192 [.138 to .309]

23. Secondary Outcome: Change in Fat Mass Ratio as Measured by DEXA Scan, in the Same Subgroup of up to 40 Participants (as in Aim 8), From Baseline to Week 96 of Treatment With Etravirine and Fixed-dose Tenofovir/Emtricitabine
Description: as for outcome 21
Time Frame: Baseline to 96 weeks
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: ratio of trunk fat % : lower limb fat %
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 25
ratio of trunk fat % : lower limb fat % | 0.06 [0.02 to 0.09]

24. Secondary Outcome: Population Pharmacokinetics of Etravirine 400 mg Once Daily, in Combination With Fixed-dose Emtricitabine-tenofovir Among Treatment-naïve HIV-1 Infected Adults
Description: Population pharmacokinetics were calculated using sparse sampling. Plasma concentrations of etravirine measured in samples from participants who provided blood samples at multiple study visits, with variation in sampling times relative to dosing of etravirine used to cover the spectrum of the dosing schedule. Model simulations and fitting were performed with NONMEM ® 7.3. (ICON, plc) and model exploration was performed with Berkeley Madonna (Berkeley, CA, USA)
Time Frame: At or after 4 weeks
Population: 57 participants who provided samples at multiple time points relative to etravirine dosing.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 57
ng/mL
  Etravirine trough plasma concentration | 217.47 [154.29 to 295.31]
  Etravirine peak plasma concentration | 480.99 [416.77 to 559.49]

25. Secondary Outcome: Population Pharmacokinetics of Etravirine 400 mg Once Daily, in Combination With Fixed-dose Emtricitabine-tenofovir Among Treatment-naïve HIV-1 Infected Adults: Etravirine AUC-24 Hours at Steady State
Description: as for outcome 24
Time Frame: At or after 4 weeks
Population: 57 participants who provided samples at multiple time points relative to etravirine dosing.
Measure: Median (Inter-Quartile Range); unit: ng*hr/mL
Arm/Group | Etravirine 400 mg Once Daily
Number analyzed (Participants) | 57
ng*hr/mL | 8024.40 [6410.20 to 9968.28]

ADVERSE EVENTS:
Time Frame: Up to 96 weeks for each participant
Description: Participants were assessed for adverse events routinely every 4 weeks in first 3 months and every 12 weeks thereafter, by standardized interview & clinical/lab exam. Labs, rash & central nervous system symptoms Grade 2 or above, other symptoms above Grade 2, and any symptom that led to change in study treatment were recorded in the database.
Arm/Group | Etravirine 400 mg Once Daily
Serious Adverse Events (participants affected / at risk) | 12/79
Other Adverse Events (participants affected / at risk) | 17/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etravirine 400 mg Once Daily (N=79)
Vomiting (Gastrointestinal disorders) | 1 (2) — Participant had longstanding history of intermittent vomiting prior to study enrollment that fluctuated while on study. He was hospitalized and stopped study drugs since the possibility that drugs were contributing to vomiting could not be excluded.
Viral gastroenteritis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) — Participant on ACE inhibitor therapy for treatment of hypertension developed renal insufficiency and hyperkalemia, resolved when ACE inhibitor discontinued.
Meningitis (Nervous system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Osteoplasty of the mandible (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 1 (1)
Disseminated atypical mycobacterium infection (Infections and infestations) | 1 (1)
malignant melanoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Skin lesion present prior to study enrollment, subsequent biopsy revealed squamous cell carcinoma.
Depressive disorder (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etravirine 400 mg Once Daily (N=79)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Elevated level of transaminase (Hepatobiliary disorders) | 9 (13) — One participant was diagnosed with acute hepatitis C at the time of transaminase elevation and was consequently discontinued from the study.
Hyperbilirubinemia (Hepatobiliary disorders) | 6 (20) — For two participants hyperbilirubinemia occurred after stopping study drug and starting other antiretrovirals due to virologic failure. One participant had sickle cell disease and elevated indirect bilirubin at entry and subsequent visits.
Neutropenia (Blood and lymphatic system disorders) | 4 (8)
Fatigue (General disorders) | 4 (4)
vomiting (Gastrointestinal disorders) | 4 (4)
Headache (General disorders) | 4 (4)
Hyperglycemia (Endocrine disorders) | 4 (7)
Hyperlipidemia (Metabolism and nutrition disorders) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes